CLINICAL TRIAL: NCT03153228
Title: The Comparison of Biomarkers of Acute Response to Cigarette Smoking and E-cigarettes Smoking Assesed in Exhaled Breath Condensate in Healthy Smokers of Traditional and Electronical Cigarettes.
Brief Title: Acute Response to Cigarette and E-cigarette Smoking Assesed in Exhaled Breath Condensate in Healthy Smokers of Traditional and E-cigarettes
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Other Study IDs: IPU-DIMPA-WUM13(2)
Record Dates: First submitted 2017-05-12; First posted 2017-05-15 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: E-cigarettes
Keywords: E-cigarettes
MeSH Terms: conditions — Vaping

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — exhaled breath condensate
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Smokers of traditional cigarettes: 29 healthy smokers of traditional cigarettes (min. 1 packyear)
- Smokers of e-cigarettes: 29 healthy smokers of e-cigarettes (min. 1 packyear)
- Control: 29 healthy volunteers.

SUMMARY:
Electronical cigarettes, also known as "e-cigarettes" are a new phenomenon, which steadily wins more aprobation among smokers. However, there exists no much data concerning the effects of acute exposure to electronic cigarettes vapour on the respiratory system.

The aim of the present study is to evaluate and compare the acute response to electronic and traditional cigarettes in healthy smokers.

DETAILED DESCRIPTION:
The aim of the study is:

* to evaluate the acute response to traditional cigarettes on the respiratory system
* to evaluate the acute response to electronic cigarettes on the respiratory system
* to assess the relationship between the type of smoked cigarettes (traditional vs. electronic) and concentration of markers of airway inflammation released in healthy smokers

Material and methods:

* 29 healthy smokers of traditional cigarettes
* 29 healthy smokers of electronic cigarettes
* 29 healthy, nonsmoking volunteers

After 8 hours of smoking abstinence:

* the spirometry test
* the first collection of the exhaled breath condensate (EBC I)
* smoking a traditional / electronic cigarette
* the second collection of the exhaled breath condensate (EBC II) - one hour after smoking
* the third collection of the exhaled breath condensate (EBC III) - six hours after smoking
* the measurement of biomarkers of oxidative stress in the EBC (isoprostane-8, malondialdehyde MDA, IL-8) and pH of the EBC

ELIGIBILITY:
Inclusion Criteria:

* healthy smokers of traditional cigarettes - min. 1 packyear
* healthy smokers of e-cigarettes - min. 1 year of smoking history
* control group - healthy nonsmoking volunteers without any history of lung disease

Exclusion Criteria:

* age below 18 years
* inhaled corticosteroid therapy at least 6 weeks prior to study enrollment
* any co-morbidities
* respiratory infections at least 6 weeks prior to study enrollment

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy smokers of traditional cigarettes, healthy smokers of e-cigarettes, healthy nonsmoking volunteers
Sampling Method: Probability Sample
Enrollment: 87 (Estimated)
Dates: Start 2017-05-08 (Actual); Primary Completion 2018-07 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Inflammatory markers in exhaled breath condensate | Approximately 1-2 months after completion of study procedures in all patients
  Inflammatory markers in exhaled breath condensate in healthy subjects, smokers of traditional cigarettes and e-cigarette smokers

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Warsaw, Banacha Hospital, Warsaw, Poland